CLINICAL TRIAL: NCT01136980
Title: A Randomized Controlled Trial Comparing Transoral Incisionless Fundoplication (TIF) Using EsophyX With Sham Procedure for the Treatment of PPI Dependent GERD Compared With Sham and Placebo Controls
Brief Title: Randomized EsophyX Versus Sham / Placebo Controlled TIF Trial: The RESPECT Study
Acronym: RESPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D01010
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Gastroesophageal Reflux Disease; Hiatal Hernia
Keywords: GERD; Esophagitis; Fundoplication; Anti-reflux surgery; PPI dependent
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal; Esophagitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham placebo procedure (Placebo Comparator): Sham Procedure: SHAM/PPI's An upper GI Endoscopy is performed with a standard endoscope, during 30-45 minutes. The patient is under general anesthesia. EGD explores the esophagus, the stomach, and the GEJ.
  Interventions: Other: Sham placebo procedure
- TIF Transoral Fundoplication (Active Comparator): Intervention: TIF 2.0/Placebo TIF Transoral Incisionless Fundoplication: A fundoplication of 270 degrees and 3cm in length was created. The EsophyX device is introduced over a standard endoscope, through the mouth, into the stomach.
  Interventions: Device: TIF Transoral Fundoplication

INTERVENTIONS:
Device: TIF Transoral Fundoplication — A novel surgical technique that creates a gastric fundoplication and restores competency of the gastroesophageal valve now exists for patients who have limited anatomic defects (small hiatal hernia). This technique is performed transorally using the EsophyX device (EndoGastric Solutions, Inc. Redmond, WA, USA) recreates a gastric fundoplication at the gastroesophageal junction by creating a flap valve at the intersection of the stomach and the esophagus by deploying polypropylene SerosaFuse fasteners (EndoGastric Solutions)
  Other Names: TIF
  Arms: TIF Transoral Fundoplication
Other: Sham placebo procedure — The Sham Procedure (control) will consist of an upper GI endoscopy that will be conducted under general anesthesia in an operating room. The surgical team will follow the same steps before, during, and after the sham procedure similar to the TIF procedure, except they will never insert the EsophyX device into the patient. The endoscope will be manipulated for 30-45 min as if the device were around it to simulate the effect of many rotations and manipulations on the esophagus.
  Other Names: Sham Procedure
  Arms: Sham placebo procedure

SUMMARY:
The objective of the study is to evaluate the relative merits, safety and effectiveness of the EsophyX transoral device in performing an advanced TIF procedure in patients with "troublesome symptoms" as defined by the Montreal consensus definition while on PPIs compared with sham and placebo controls.

DETAILED DESCRIPTION:
Primary Effectiveness Endpoint: A clinically significant reduction in GERD symptoms, specifically "Troublesome" regurgitation with or without heartburn assessed by the Reflux Disease Questionnaire (RDQ).

Troublesome symptoms are those which occur a minimum of 2 days a week and are at least moderate in severity.

Secondary Effectiveness Endpoint: The normalization of esophageal acid exposure at 6 months and a clinically significant reduction in PPI usage at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Dependent upon daily PPIs for > 6 months
* Troublesome symptoms, specifically heartburn or regurgitation, while on 40 mg of omeprazole or equivalent.

Troublesome heartburn or regurgitation symptoms are those which occur a minimum of 2-3 days a week and are at least moderate in severity.

* Abnormal ambulatory pH study off PPI therapy for 7 days.
* Normal or near normal esophageal motility (by manometry)
* Hiatal hernia axial height is no larger than 2 cm and the transverse dimension should not exceed 2.5 cm
* Patient willing to cooperate with post-operative dietary recommendations and assessment tests
* Signed informed consent

Exclusion Criteria:

* BMI > 35
* Hiatal hernia > 2 cm
* Esophagitis Los Angeles grade C or D
* Esophageal ulcer
* Esophageal stricture
* Esophageal motility disorder
* Pregnancy or plans for pregnancy in the next 12 months (in females)
* Immunosuppression
* ASA > 2
* Portal hypertension and/or varices
* History of previous resective gastric or esophageal surgery, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, or cirrhosis
* Active gastro-duodenal ulcer disease
* Gastric outlet obstruction or stenosis
* Severe gastroparesis or delayed gastric emptying confirmed by solid-phase gastric emptying study if patient complains of postprandial satiety during assessment
* Coagulation disorders
* Interprocedural determination of anatomical presentation which in the opinion of the surgeon does not allow safe device introduction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hunter, MD FACS, Principal Investigator — Oregon Health and Science University
Locations (9):
- United States (9):
  - Cedars Sinai Medical Center, Los Angeles, California
  - SurgOne PC, Englewood, Colorado
  - Northwestern University, Chicago, Illinois
  - Ohio State University Hospital, Columbus, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas, Health Science Center at Houston, Houston, Texas
  - Reston Surgical Associates, Reston, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hunter JG, Kahrilas PJ, Bell RC, Wilson EB, Trad KS, Dolan JP, Perry KA, Oelschlager BK, Soper NJ, Snyder BE, Burch MA, Melvin WS, Reavis KM, Turgeon DG, Hungness ES, Diggs BS. Efficacy of transoral fundoplication vs omeprazole for treatment of regurgitation in a randomized controlled trial. Gastroenterology. 2015 Feb;148(2):324-333.e5. doi: 10.1053/j.gastro.2014.10.009. Epub 2014 Oct 13. PMID 25448925

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Placebo Procedure | TIF Transoral Fundoplication
Started | 42 | 87
Completed | 28 | 76
Not Completed | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Placebo Procedure | TIF Transoral Fundoplication | Total
Number analyzed (Participants) | 42 | 87 | 129
Age, Continuous [Median (Full Range); unit: years] | 55 [22 to 73] | 52 [22 to 74] | 53 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 40 | 66
  Male | 16 | 47 | 63
Region of Enrollment [Number; unit: participants]
  United States | 42 | 87 | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinically Significant Reduction in Gastroesophageal Reflux Disease (GERD) Symptoms (Specifically "Troublesome" Regurgitation With or Without Heartburn as Assessed by the RDQ Per the Montreal Consensus Definition,
Description: Primary efficacy Hypothesis 1: At 6-month follow-up, the proportion of Transesophageal Incisionless Fundoplication (TIF)2+Placebo pts who are free of "troublesome" symptoms will be statistically significantly larger than those randomized to the Sham+PPI (Proton Pump Inhibitor) treatment group.
Time Frame: 6 month follow up
Population: Patients completing 6 month post-procedure follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Placebo Procedure | TIF Transoral Fundoplication
Number analyzed (Participants) | 28 | 76
Participants | 17 | 54
Statistical Analysis 1: Comparison: Sham Placebo Procedure vs TIF Transoral Fundoplication; Test type: Superiority; p < 0.028, Chi-squared

2. Secondary Outcome: Normalization of Esophageal Acid Exposure - as Measured by DeMeester Score
Description: DeMeester Score is a composite score taking into consideration reflux episodes, percentage of time pH is < 4 and others. DMS was first reported in 1974 by Johnson and DeMeester. It is a composite score that measures acid exposure during prolonged ambulatory pH monitoring. The parameters that constitute the score are:
  1. total number of episodes of reflux, - reflux is undesirable, therefore lower numbers are better, higher numbers are worse. Ideally there would be zero reflux episodes.
  2. % total time esophageal pH < 4, upright position and supine position, respectively - pH < 4 is undesirable, therefor lower percentages are better
  3. number of episodes longer than 5 minutes, - lower is better
  4. maximal reflux duration, (reflux is undesirable - lower is better
  5. total percentage of time with pH below 4 - below 4 is undesirable - lower is better
  The composite score can be obtained by adding the scores calculated for each of the six components.
Time Frame: 6 months post procedure
Population: Patients that completed 6 month follow-up. NOTE: greater than 14.72 is considered abnormal, 14.72-50 is regarded as mild GERD, 51-100 is regarded as moderate GERD, and greater than 100 is regarded as severe GERD.
Measure: Mean (Full Range); unit: Composite DeMeester Score
Arm/Group | Sham Placebo Procedure | TIF Transoral Fundoplication
Number analyzed (Participants) | 28 | 76
Composite DeMeester Score
  Pre-Procedure DeMeester Score | 30.9 [14 to 50] | 33.6 [14 to 110]
  6 month post-procedure DeMeester Score | 32.7 [1 to 65] | 23.9 [0 to 80]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sham Placebo Procedure | TIF Transoral Fundoplication
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/87
Serious Adverse Events (participants affected / at risk) | 1/42 | 3/87
Other Adverse Events (participants affected / at risk) | 0/42 | 4/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Placebo Procedure (N=42) | TIF Transoral Fundoplication (N=87)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Temporary epigastric /abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Placebo Procedure (N=42) | TIF Transoral Fundoplication (N=87)
Temporary epigastric / abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Intent to treat (ITT) analysis included 12 patients with limited follow-up data. Assessment of the primary end point at 6 months can be viewed as premature by some; however, we believed it likely that delaying the primary end point beyond 6 months would risk patients not entering or dropping out of the study prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No